CLINICAL TRIAL: NCT04447040
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate Five Strengths of a Fixed Combination of Acetaminophen/Naproxen Sodium in Postoperative Dental Pain
Brief Title: Acetaminophen/Naproxen Sodium Dose Ranging Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Consumer Inc., McNeil Consumer Healthcare Division (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCSPAA002398
Record Dates: First submitted 2020-06-23; First posted 2020-06-25 (Actual); Results first posted 2024-04-11 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2024-03

CONDITIONS: Pain
Keywords: Analgesics; Dental Pain; Acetaminophen; Naproxen Sodium; Pain; Fixed-Dose
MeSH Terms: conditions — Pain; Toothache | interventions — Acetaminophen

STUDY DESIGN:
Intervention Model Description: Post-operative dental pain following third molar extraction.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Acetaminophen/naproxen sodium Dose A (Experimental): Acetaminophen/naproxen sodium Dose A administered as a single two-tablet dose.
  Interventions: Drug: Acetaminophen/naproxen sodium Dose A
- Acetaminophen/naproxen sodium Dose B (Experimental): Acetaminophen/naproxen sodium Dose B administered as a single two-tablet dose.
  Interventions: Drug: Acetaminophen/naproxen sodium Dose B
- Acetaminophen/naproxen sodium Dose C (Experimental): Acetaminophen/naproxen sodium Dose C administered as a single two-tablet dose.
  Interventions: Drug: Acetaminophen/naproxen sodium Dose C
- Acetaminophen/naproxen sodium Dose D (Experimental): Acetaminophen/naproxen sodium Dose D administered as a single two-tablet dose.
  Interventions: Drug: Acetaminophen/naproxen sodium Dose D
- Acetaminophen/naproxen sodium Dose E (Experimental): Acetaminophen/naproxen sodium Dose E administered as a single two-tablet dose.
  Interventions: Drug: Acetaminophen/naproxen sodium Dose E
- Placebo (Placebo Comparator): Placebo tablets administered as a single two-tablet dose.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetaminophen/naproxen sodium Dose A — Acetaminophen/naproxen sodium Dose A administered as a single two-tablet dose.
  Arms: Acetaminophen/naproxen sodium Dose A
Drug: Acetaminophen/naproxen sodium Dose B — Acetaminophen/naproxen sodium Dose B administered as a single two-tablet dose.
  Arms: Acetaminophen/naproxen sodium Dose B
Drug: Acetaminophen/naproxen sodium Dose C — Acetaminophen/naproxen sodium Dose C administered as a single two-tablet dose.
  Arms: Acetaminophen/naproxen sodium Dose C
Drug: Acetaminophen/naproxen sodium Dose D — Acetaminophen/naproxen sodium Dose D administered as a single two-tablet dose.
  Arms: Acetaminophen/naproxen sodium Dose D
Drug: Acetaminophen/naproxen sodium Dose E — Acetaminophen/naproxen sodium Dose E administered as a single two-tablet dose.
  Arms: Acetaminophen/naproxen sodium Dose E
Drug: Placebo — Placebo tablets administered as a single two-tablet dose.
  Arms: Placebo

SUMMARY:
Study assessing the relative efficacy of five strengths of a fixed combination of acetaminophen and naproxen sodium is being investigated to help inform selection of dose(s) for further development and to evaluate the safety of a fixed combination of naproxen sodium and acetaminophen.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study to evaluate the analgesic efficacy and safety profile of the following doses of a fixed combination of Acetaminophen (APAP)/Naproxen sodium (NPX) administered as a single two-tablet dose:[Acetaminophen/Naproxen Sodium Dose A, Acetaminophen/Naproxen Sodium Dose B, Acetaminophen/Naproxen Sodium Dose C, Acetaminophen/Naproxen Sodium Dose D, Acetaminophen/Naproxen Sodium Dose E and Placebo] following surgical extraction of four third molars.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females 17-50 years old
2. Weigh 100 pounds or greater and have a body mass index (BMI) of 17.5-35.4 (inclusive) at screening
3. Surgical removal of three or four third molars, of which, two must be mandibular impactions
4. Meets requirements for post-surgical pain level
5. Females of childbearing potential and males agree to contraceptive requirements of study
6. Have a negative urine drug screen at screening, and on day of surgical procedure

Exclusion Criteria:

1. Pregnant female, breastfeeding, trying to become pregnant or male with pregnant partner or partner currently trying to become pregnant
2. Have a known allergy or hypersensitivity to naproxen or other NSAIDs, including aspirin, or to acetaminophen, oxycodone or other opioids;
3. Not able to swallow whole large tablets or capsules
4. History of any condition (s) in investigator's opinion, may jeopardize subject safety, well-being and integrity of study
5. Use analgesics 5 or more times per week
6. History of chronic tranquilizer use, heavy drinking, or substance abuse, as judged by the investigator site staff, in the last 5 years
7. Use of any immunosuppressive drugs within 2 weeks of screening
8. History of endoscopically documented peptic ulcer disease or bleeding disorder in the last 2 years

Ages: 17 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 304 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2021-04-09 (Actual); Study Completion 2021-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd Bertoch, MD, Principal Investigator — JBR Clinical Research
Locations (1):
- JBR Clinical Research, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Consumer Inc. has an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu.

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants who underwent dental extraction of three or four third molars received a single oral dose of two placebo tablets on Day 1 post dental extraction.
- Acetaminophen/Naproxen Sodium Dose A: Participants who underwent dental extraction of three or four third molars received two tablets of fixed combination of acetaminophen and naproxen sodium Dose A orally on Day 1 post dental extraction.
- Acetaminophen/Naproxen Sodium Dose B: Participants who underwent dental extraction of three or four third molars received two tablets of fixed combination of acetaminophen and naproxen sodium Dose B orally on Day 1 post dental extraction.
- Acetaminophen/Naproxen Sodium Dose C: Participants who underwent dental extraction of three or four third molars received two tablets of fixed combination of acetaminophen and naproxen sodium Dose C orally on Day 1 post dental extraction.
- Acetaminophen/Naproxen Sodium Dose D: Participants who underwent dental extraction of three or four third molars received two tablets of fixed combination of acetaminophen and naproxen sodium Dose D orally on Day 1 post dental extraction.
- Acetaminophen/Naproxen Sodium Dose E: Participants who underwent dental extraction of three or four third molars received two tablets of fixed combination of acetaminophen and naproxen sodium Dose E orally on Day 1 post dental extraction.
Period: Overall Study
Arm/Group | Placebo | Acetaminophen/Naproxen Sodium Dose A | Acetaminophen/Naproxen Sodium Dose B | Acetaminophen/Naproxen Sodium Dose C | Acetaminophen/Naproxen Sodium Dose D | Acetaminophen/Naproxen Sodium Dose E
Started | 53 | 49 | 53 | 52 | 51 | 46
Completed | 51 | 47 | 49 | 48 | 50 | 43
Not Completed | 2 | 2 | 4 | 4 | 1 | 3
Not completed — Lost to Follow-up | 2 | 1 | 3 | 3 | 1 | 3
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Acetaminophen/Naproxen Sodium Dose A | Acetaminophen/Naproxen Sodium Dose B | Acetaminophen/Naproxen Sodium Dose C | Acetaminophen/Naproxen Sodium Dose D | Acetaminophen/Naproxen Sodium Dose E | Total
Number analyzed (Participants) | 53 | 49 | 53 | 52 | 51 | 46 | 304
Age, Continuous [Mean (Standard Deviation); unit: Years] | 18.5 (1.78) | 18.4 (1.83) | 18.6 (2.05) | 18.7 (1.95) | 18.5 (1.82) | 18.2 (1.50) | 18.5 (1.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 27 | 26 | 25 | 27 | 24 | 154
  Male | 28 | 22 | 27 | 27 | 24 | 22 | 150
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 6 | 5 | 2 | 2 | 9 | 36
  Not Hispanic or Latino | 40 | 43 | 48 | 50 | 49 | 37 | 267
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Asian | 1 | 1 | 1 | 2 | 1 | 1 | 7
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 1 | 0 | 0 | 3
  Black or African American | 1 | 0 | 0 | 0 | 0 | 0 | 1
  White | 50 | 48 | 51 | 48 | 50 | 45 | 292
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Time Weighted Sum of Pain Intensity Difference Score From Baseline (0 Hour) to 12 Hours (SPID 0-12)
Description: Time weighted sum of the pain intensity difference (SPID) score is derived from pain intensity difference (PID) score. Pain intensity-numerical rating scale (PI-NRS) was used to assess pain intensity on scale ranged from 0 (no pain) to 10 (very severe pain), higher score indicated severe pain intensity. PID score was the difference between baseline pain intensity and pain intensity at assessment timepoint (12 hours). The SPID scores were derived by first multiplying each PID score by the time from the previous time point and adding these time weighted PID scores together over the interval from 0 to 12 hours. The possible range of SPID for 0 to 12 hours was from -120 to 120. A higher value of SPID indicated greater pain relief.
Time Frame: Baseline (0 hour) up to 12 hours post-dose on Day 1
Population: Intent-to-Treat (ITT) analysis set included all randomized participants.
Measure: Least Squares Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Acetaminophen/Naproxen Sodium Dose A | Acetaminophen/Naproxen Sodium Dose B | Acetaminophen/Naproxen Sodium Dose C | Acetaminophen/Naproxen Sodium Dose D | Acetaminophen/Naproxen Sodium Dose E
Number analyzed (Participants) | 53 | 49 | 53 | 52 | 51 | 46
Units on a scale | 5.59 (3.741) | 37.08 (3.892) | 46.98 (3.740) | 52.45 (3.779) | 59.63 (3.813) | 65.52 (4.027)
Statistical Analysis 1: Comparison: Placebo vs Acetaminophen/Naproxen Sodium Dose A; Test type: Superiority; p < 0.001, ANOVA; Least square (LS) Mean Difference = 31.48, 95% CI 2-sided [20.90 to 42.07], Standard Error of Mean 5.379
Statistical Analysis 2: Comparison: Placebo vs Acetaminophen/Naproxen Sodium Dose B; Test type: Superiority; p < 0.001, ANOVA; LS Mean Difference = 41.38, 95% CI 2-sided [31.02 to 51.75], Standard Error of Mean 5.267
Statistical Analysis 3: Comparison: Placebo vs Acetaminophen/Naproxen Sodium Dose C; Test type: Superiority; p < 0.001, ANOVA; LS Mean Difference = 46.86, 95% CI 2-sided [36.44 to 57.27], Standard Error of Mean 5.292
Statistical Analysis 4: Comparison: Placebo vs Acetaminophen/Naproxen Sodium Dose D; Test type: Superiority; p < 0.001, ANOVA; LS Mean Difference = 54.04, 95% CI 2-sided [43.57 to 64.51], Standard Error of Mean 5.321
Statistical Analysis 5: Comparison: Placebo vs Acetaminophen/Naproxen Sodium Dose E; Test type: Superiority; p < 0.001, ANOVA; LS Mean Difference = 59.92, 95% CI 2-sided [49.16 to 70.68], Standard Error of Mean 5.468

2. Secondary Outcome: Time Weighted Sum of Total Pain Relief Score From Baseline (0 Hour) to 12 Hours (TOTPAR 0-12)
Description: Time weighted total pain relief (TOTPAR) was measured using a Pain Relief Numerical Rating Scale (PR-NRS) ranging from 0 to10 (0 = no relief, 10 = complete relief). A higher score indicated greater pain relief. Total pain relief scores (TOTPARs) were calculated by multiplying the pain relief score at each post-dose time point by the duration (in hours) since the preceding time point and then summing these values. The minimum value was 0, and the maximum value was 120. Higher scores were indicative of more pain relief.
Time Frame: Baseline (0 hour) up to 12 hours post-dose on Day 1
Population: ITT analysis set included all randomized participants.
Measure: Least Squares Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Acetaminophen/Naproxen Sodium Dose A | Acetaminophen/Naproxen Sodium Dose B | Acetaminophen/Naproxen Sodium Dose C | Acetaminophen/Naproxen Sodium Dose D | Acetaminophen/Naproxen Sodium Dose E
Number analyzed (Participants) | 53 | 49 | 53 | 52 | 51 | 46
Units on a scale | 18.40 (4.550) | 54.06 (4.734) | 67.45 (4.548) | 72.04 (4.597) | 79.33 (4.637) | 85.98 (4.898)
Statistical Analysis 1: Comparison: Placebo vs Acetaminophen/Naproxen Sodium Dose A; Test type: Superiority; p < 0.001, ANOVA; LS Mean Difference = 35.66, 95% CI 2-sided [22.79 to 48.54], Standard Error of Mean 6.542
Statistical Analysis 2: Comparison: Placebo vs Acetaminophen/Naproxen Sodium Dose B; Test type: Superiority; p < 0.001, ANOVA; LS Mean Difference = 49.04, 95% CI 2-sided [36.44 to 61.65], Standard Error of Mean 6.407
Statistical Analysis 3: Comparison: Placebo vs Acetaminophen/Naproxen Sodium Dose C; Test type: Superiority; p < 0.001, ANOVA; LS Mean Difference = 53.64, 95% CI 2-sided [40.97 to 66.31], Standard Error of Mean 6.437
Statistical Analysis 4: Comparison: Placebo vs Acetaminophen/Naproxen Sodium Dose D; Test type: Superiority; p < 0.001, ANOVA; LS Mean Difference = 60.93, 95% CI 2-sided [48.19 to 73.67], Standard Error of Mean 6.472
Statistical Analysis 5: Comparison: Placebo vs Acetaminophen/Naproxen Sodium Dose E; Test type: Superiority; p < 0.001, ANOVA; LS Mean Difference = 67.58, 95% CI 2-sided [54.49 to 80.67], Standard Error of Mean 6.650

3. Secondary Outcome: Time Weighted Sum of Pain Intensity Difference Score From 6 Hours to 12 Hours (SPID 6-12)
Description: Time weighted sum of the pain intensity difference (SPID) score is derived from PID score. PI-NRS was used to assess pain intensity on scale ranged from 0 (no pain) to 10 (very severe pain), higher score indicated severe pain intensity. PID was the difference between pain intensity at 6 hours and pain intensity at assessment timepoint (12 hours). The SPID scores were derived by first multiplying each PID score by the time from the previous time point and adding these time weighted PID scores together over the intervals from 6 to 12 hours (6 hours). The possible range of SPID for 6 to12 hours was from -60 to 60. A higher value of SPID indicated greater pain relief.
Time Frame: From 6 hours up to 12 hours post-dose on Day 1
Population: ITT analysis set included all randomized participants.
Measure: Least Squares Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Acetaminophen/Naproxen Sodium Dose A | Acetaminophen/Naproxen Sodium Dose B | Acetaminophen/Naproxen Sodium Dose C | Acetaminophen/Naproxen Sodium Dose D | Acetaminophen/Naproxen Sodium Dose E
Number analyzed (Participants) | 53 | 49 | 53 | 52 | 51 | 46
Units on a scale | 2.58 (2.154) | 15.12 (2.241) | 20.31 (2.153) | 24.47 (2.176) | 27.59 (2.195) | 31.89 (2.318)
Statistical Analysis 1: Comparison: Placebo vs Acetaminophen/Naproxen Sodium Dose A; Test type: Superiority; p < 0.001, ANOVA; LS mean Difference = 12.53, 95% CI 2-sided [6.44 to 18.63], Standard Error of Mean 3.097
Statistical Analysis 2: Comparison: Placebo vs Acetaminophen/Naproxen Sodium Dose B; Test type: Superiority; p < 0.001, ANOVA; LS MEAN Difference = 17.73, 95% CI 2-sided [11.76 to 23.70], Standard Error of Mean 3.032
Statistical Analysis 3: Comparison: Placebo vs Acetaminophen/Naproxen Sodium Dose C; Test type: Superiority; p < 0.001, ANOVA; LS Mean Difference = 21.88, 95% CI 2-sided [15.89 to 27.88], Standard Error of Mean 3.047
Statistical Analysis 4: Comparison: Placebo vs Acetaminophen/Naproxen Sodium Dose D; Test type: Superiority; p < 0.001, ANOVA; LS Mean Difference = 25.01, 95% CI 2-sided [18.98 to 31.03], Standard Error of Mean 3.063
Statistical Analysis 5: Comparison: Placebo vs Acetaminophen/Naproxen Sodium Dose E; Test type: Superiority; p < 0.001, ANOVA; LS Mean Difference = 29.30, 95% CI 2-sided [23.11 to 35.50], Standard Error of Mean 3.148

4. Secondary Outcome: Time to First Use of Rescue Analgesic Medication
Description: Time to first use of rescue analgesic medication was measured as the elapsed time (in minutes) from when the investigational product was given until the time rescue analgesic was first given. Participants who did not use rescue medication during the 24 hour study period had their time to rescue set to 24 hours and were censored at 24 hours. Kaplan-Meier method was used for the analysis.
Time Frame: From 0 minute up to 1440 minutes post-dose (that is, up to 24 hours post-dose) on Day 1
Population: ITT analysis set included all randomized participants.
Measure: Median (Full Range); unit: Minutes
Arm/Group | Placebo | Acetaminophen/Naproxen Sodium Dose A | Acetaminophen/Naproxen Sodium Dose B | Acetaminophen/Naproxen Sodium Dose C | Acetaminophen/Naproxen Sodium Dose D | Acetaminophen/Naproxen Sodium Dose E
Number analyzed (Participants) | 53 | 49 | 53 | 52 | 51 | 46
Minutes | 90.0 [38 to 1440] | 898.0 [33 to 1440] | 1195.0 [30 to 1440] | NA [0 to 1440] — Median was not estimable because fewer than 50% of participants required rescue medication. | NA [68 to 1440] — Median was not estimable because fewer than 50% of participants required rescue medication. | NA [497 to 1440] — Median was not estimable because fewer than 50% of participants required rescue medication.
Statistical Analysis 1: Comparison: Placebo vs Acetaminophen/Naproxen Sodium Dose A; Test type: Superiority; p < 0.001, Wilcoxon test
Statistical Analysis 2: Comparison: Placebo vs Acetaminophen/Naproxen Sodium Dose B; Test type: Superiority; p < 0.001, Wilcoxon test
Statistical Analysis 3: Comparison: Placebo vs Acetaminophen/Naproxen Sodium Dose C; Test type: Superiority; p < 0.001, Wilcoxon test
Statistical Analysis 4: Comparison: Placebo vs Acetaminophen/Naproxen Sodium Dose D; Test type: Superiority; p < 0.001, Wilcoxon test
Statistical Analysis 5: Comparison: Placebo vs Acetaminophen/Naproxen Sodium Dose E; Test type: Superiority; p < 0.001, Wilcoxon test

5. Secondary Outcome: Proportion of Participants Who Required Rescue Analgesic Medication
Description: Proportion (cumulative data) of participants who used rescue analgesic medication through 24 hours post study drug administration on Day 1 which was assessed by using Kaplan-Meier estimates were reported.
Time Frame: From 0 hour up to 24 hours post-dose on Day 1
Population: ITT analysis set included all randomized participants.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Placebo | Acetaminophen/Naproxen Sodium Dose A | Acetaminophen/Naproxen Sodium Dose B | Acetaminophen/Naproxen Sodium Dose C | Acetaminophen/Naproxen Sodium Dose D | Acetaminophen/Naproxen Sodium Dose E
Number analyzed (Participants) | 53 | 49 | 53 | 52 | 51 | 46
Proportion of participants | 0.792 [0.675 to 0.889] | 0.571 [0.439 to 0.711] | 0.519 [0.392 to 0.659] | 0.353 [0.239 to 0.500] | 0.353 [0.239 to 0.500] | 0.152 [0.076 to 0.293]
Statistical Analysis 1: Comparison: Placebo vs Acetaminophen/Naproxen Sodium Dose A; Test type: Superiority; p = 0.014, Wald method
Statistical Analysis 2: Comparison: Placebo vs Acetaminophen/Naproxen Sodium Dose B; Test type: Superiority; p = 0.002, Wald method
Statistical Analysis 3: Comparison: Placebo vs Acetaminophen/Naproxen Sodium Dose C; Test type: Superiority; p < 0.001, Wald method
Statistical Analysis 4: Comparison: Placebo vs Acetaminophen/Naproxen Sodium Dose D; Test type: Superiority; p < 0.001, Wald method
Statistical Analysis 5: Comparison: Placebo vs Acetaminophen/Naproxen Sodium Dose E; Test type: Superiority; p < 0.001, Wald method

ADVERSE EVENTS:
Time Frame: From baseline (Day 1; day of surgery) up to Day 10
Description: The safety analysis set included all participants who were randomized and took investigational product. Analyzed based on the actual received treatment.
Arm/Group | Placebo | Acetaminophen/Naproxen Sodium Dose A | Acetaminophen/Naproxen Sodium Dose B | Acetaminophen/Naproxen Sodium Dose C | Acetaminophen/Naproxen Sodium Dose D | Acetaminophen/Naproxen Sodium Dose E
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/49 | 0/53 | 0/52 | 0/51 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/49 | 0/53 | 0/52 | 0/51 | 0/46
Other Adverse Events (participants affected / at risk) | 12/53 | 7/49 | 6/53 | 5/52 | 3/51 | 3/46
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=53) | Acetaminophen/Naproxen Sodium Dose A (N=49) | Acetaminophen/Naproxen Sodium Dose B (N=53) | Acetaminophen/Naproxen Sodium Dose C (N=52) | Acetaminophen/Naproxen Sodium Dose D (N=51) | Acetaminophen/Naproxen Sodium Dose E (N=46)
Nausea (Gastrointestinal disorders) | 9 | 5 | 2 | 2 | 2 | 1
Vomiting (Gastrointestinal disorders) | 6 | 1 | 2 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 1 | 1 | 0 | 0 | 2
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0
Alveolar osteitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Corona virus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 1 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of study results by the Investigator is discussed in the Clinical Study Agreement, as appropriate. Results from this study may be published in the form of oral or written presentations at scientific meetings or as one or more peer-reviewed journal articles. In these cases, no information on individual subjects will be revealed.

DOCUMENTS (2):
  • Study Protocol (2020-11-25): https://cdn.clinicaltrials.gov/large-docs/40/NCT04447040/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-17): https://cdn.clinicaltrials.gov/large-docs/40/NCT04447040/SAP_001.pdf